CLINICAL TRIAL: NCT07162090
Title: Observation of the Impact of Hypoxia - Inducible Factor Prolyl Hydroxylase Inhibitors on Sarcopenia in Hemodialysis Patients
Brief Title: Hypoxia-inducible Factor Prolyl Hydroxylase Inhibitors on Sarcopenia in Hemodialysis Patients
Acronym: HIF-PHI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Peng-cheng Xu, chief physician, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2025-YX-317-01
Record Dates: First submitted 2025-08-04; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Anemia Associated With Chronic Kidney Disease (CKD); Dialysis Patients
Keywords: Sarcopenia; Anemia
MeSH Terms: conditions — Sarcopenia; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving treatment with Roxadustat (Experimental): Roxadustat is administered at an initial dose of 50 mg per oral administration, three times a week. Complete blood count and serum iron levels are re - evaluated monthly. The dosage is adjusted based on the rate of increase in hemoglobin levels. Observations were made every six weeks starting from the initiation of treatment, and the entire observation period lasted for 24 weeks.
  Interventions: Drug: Roxadustat
- Patients receiving treatment with recombinant human erythropoietin (Active Comparator): For recombinant human erythropoietin, the initial dosage is 3000 international units (IU) per administration. It is administered via subcutaneous injection three times a week. The blood routine and serum iron levels are re - examined monthly. The dosage is adjusted according to the rate of increase in hemoglobin. Observations were made every six weeks starting from the initiation of treatment, and the entire observation period lasted for 24 weeks.
  Interventions: Drug: Recombinant human erythropoietin (EPO)

INTERVENTIONS:
Drug: Roxadustat — Patients were administered roxadustat orally to observe its impacts on renal anemia and sarcopenia.
  Other Names: HIF-PHI
  Arms: Patients receiving treatment with Roxadustat
Drug: Recombinant human erythropoietin (EPO) — Recombinant human erythropoietin was administered to patients as a control group to investigate its impacts on renal anemia and sarcopenia.
  Other Names: rHuEPO
  Arms: Patients receiving treatment with recombinant human erythropoietin

SUMMARY:
Sarcopenia, abbreviated as muscle loss, is a prevalent complication among patients with chronic kidney disease (CKD), particularly those with end - stage renal disease (ESRD). It significantly impacts patients' quality of life. The prevalence of sarcopenia in patients receiving maintenance hemodialysis (MHD) ranges from 32.7% to 73.5%, which is substantially higher than that in the general population (5% - 13%). Sarcopenia significantly elevates the mortality risk in MHD patients. Specifically, sarcopenia patients experience an increased all - cause mortality rate, a heightened risk of cardiovascular events, a decline in quality of life, and an augmented risk of falls and fractures. A close pathophysiological relationship exists between the hypoxia - inducible factor - 1 (HIF - 1) pathway and sarcopenia. HIF - 1α serves as a key transcription factor for cells to respond to hypoxic conditions. Under normoxic conditions, HIF - 1α is hydroxylated by prolyl hydroxylase (PHD) and subsequently undergoes ubiquitination - mediated degradation. Conversely, under hypoxic circumstances, HIF - 1α is stably expressed, translocates into the nucleus, and activates downstream target genes. HIF - 1α promotes the expression of genes associated with glycolysis, such as GLUT1 and LDHA, while inhibiting mitochondrial oxidative phosphorylation. This results in a shift of skeletal muscle energy metabolism from aerobic to anaerobic pathways. Research has revealed that the protein level of HIF - 1α is significantly decreased in sarcopenia patients. Roxadustat capsules, an oral medication, represent the world's first small - molecule hypoxia - inducible factor prolyl hydroxylase inhibitor (HIF - PHI) developed for the treatment of renal anemia. The physiological function of HIF - 1α not only enhances the expression of erythropoietin but also upregulates the expression of erythropoietin receptors and proteins involved in promoting iron absorption and circulation. Theoretically, roxadustat has the potential to improve sarcopenia. However, due to its prominent effect on anemia correction, it is currently only clinically applicable to anemic patients. This study aims to use ESA as a control to investigate the effect of roxadustat on sarcopenia in hemodialysis patients during the treatment of renal anemia.

DETAILED DESCRIPTION:
Sarcopenia, commonly abbreviated as age-related muscle loss, represents a highly prevalent and serious complication among patients suffering from chronic kidney disease (CKD), particularly those advancing to end-stage renal disease (ESRD). It profoundly undermines multiple aspects of patients' lives, leading to markedly reduced mobility, increased dependency, and overall diminished quality of life. Defined as a progressive and generalized skeletal muscle disorder, sarcopenia involves the accelerated loss of muscle mass and function, which goes beyond normal aging. Clinically, it is diagnosed through measurements showing declines in three key areas: muscle mass, muscle strength, and physical performance. Although initially recognized and characterized in the elderly, it is now evident that sarcopenia disproportionately affects individuals with chronic conditions such as CKD.

The prevalence of sarcopenia is strikingly elevated in patients undergoing maintenance hemodialysis (MHD). Studies report that between 32.7% and 73.5% of MHD patients are affected, a rate substantially higher than the 5% to 13% observed in the general population. This condition is not merely a comorbidity; it significantly increases the risk of mortality. Specifically, MHD patients with sarcopenia face higher all-cause mortality, greater susceptibility to cardiovascular events, reduced quality of life, and elevated risks of falls and fractures. Consequently, the development of effective treatments for sarcopenia is of major clinical importance for this vulnerable population.

The pathogenesis of sarcopenia in MHD patients is multifactorial. Major contributing factors include nutritional and metabolic imbalances. During hemodialysis, significant quantities of amino acids are lost, and many patients experience poor appetite, leading to chronically inadequate protein intake. Additionally, a state of chronic micro-inflammation promotes muscle protein breakdown via activation of proteolytic pathways, thereby accelerating muscle wasting. Other metabolic abnormalities-such as metabolic acidosis, insulin resistance, and vitamin D deficiency-further exacerbate the loss of muscle mass and function.

Although current management strategies focus on addressing these factors through nutritional support, exercise interventions, and metabolic corrections, the overall outcomes remain suboptimal for a significant proportion of patients. Hence, there is a pressing need to explore targeted pharmacological therapies. Recent research has shed light on the hypoxia-inducible factor-1 (HIF-1) pathway, which appears to have a close pathophysiological relationship with muscle homeostasis. HIF-1α, a central transcription factor that mediates cellular adaptation to hypoxia, is regulated by oxygen-dependent degradation. Under normal oxygen conditions, prolyl hydroxylase domain (PHD) enzymes hydroxylate HIF-1α, marking it for ubiquitination and proteasomal degradation. Under hypoxic conditions, however, HIF-1α accumulates, translocates to the nucleus, dimerizes with HIF-1β, and activates the transcription of numerous target genes.

Interestingly, HIF-1α drives the expression of genes related to glycolysis (e.g., GLUT1 and LDHA) and suppresses mitochondrial oxidative phosphorylation, shifting energy production in skeletal muscle from aerobic to anaerobic metabolism. Notably, research has shown that protein levels of HIF-1α are significantly reduced in individuals with sarcopenia, suggesting an impaired hypoxic response mechanism that may be essential for activating muscle regeneration. Therefore, therapeutic activation of HIF-1α and its target genes has emerged as a promising strategy to ameliorate skeletal muscle atrophy.

Roxadustat, an orally administered capsule, is the world's first hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI) approved for the treatment of renal anemia. Its mechanism of action involves mimicking α-ketoglutarate, thereby inhibiting PHD enzymes and stabilizing HIF-1α. This not only enhances erythropoietin (EPO) expression but also upregulates erythropoietin receptors and proteins that facilitate iron absorption and recycling. By restoring iron homeostasis and promoting erythropoiesis, roxadustat effectively corrects anemia. Beyond its primary use in renal anemia, roxadustat is now being investigated and applied in other anemia types.

Theoretical and preclinical evidence suggests that roxadustat may also confer benefits in sarcopenia. However, given its primary indication for anemia, current clinical use is restricted to anemic patients. Renal anemia is exceedingly common in hemodialysis patients, historically managed with injectable recombinant erythropoietin (erythropoiesis-stimulating agents, ESAs). While ESAs effectively raise hemoglobin levels, they are not expected to directly influence muscle mass or function. In contrast, roxadustat has demonstrated superior efficacy in correcting renal anemia compared to ESA therapy. Nonetheless, no direct comparative studies have yet evaluated the effects of roxadustat versus ESA on sarcopenia in the hemodialysis population.

Therefore, this study is designed to address the existing gap by utilizing ESA as a control to evaluate the potential benefits of roxadustat on sarcopenia in hemodialysis patients, while concurrently targeting its intended treatment for renal anemia. The findings may offer valuable insights into a novel therapeutic approach that transcends mere anemia management and aims to enhance musculoskeletal health within this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old (inclusive), gender unrestricted.
* End-stage renal disease and maintenance hemodialysis for at least 16 weeks.
* The average Hb level is 7.0~10.0 g/dL (the last two evaluations).
* And have not received or have discontinued ESA/roxadustat treatment.
* Vascular access: internal fistula or long-term hemodialysis catheter.
* Weight between 45-100 kg.
* Sarcopenia Diagnosis (Reference: AWGS 2019 Consensus):
* Decreased muscle strength: Male grip strength < 28 kg, female grip strength < 18 kg.
* Muscle mass decline: Assessed by bioelectrical impedance analysis (BIA) or dual-energy X-ray absorptiometry (DXA), it is characterized by appendicular skeletal muscle mass index (ASMI): < 7.0 kg/m² for men and < 5.7 kg/m² for women (BIA standard, the device and formula used should be specified).
* Sarcopenia can be diagnosed when both "decreased muscle strength" and "reduced muscle mass" are present. If resources permit, "decreased physical function" (such as a 6-meter walking speed < 1.0 m/s) can be added as an indicator for severity grading.
* Voluntary participation in this study.
* Must be able to swallow tablets。

Exclusion Criteria:

* Non-renal anemia: Anemia caused by other main reasons (such as thalassemia, megaloblastic anemia due to vitamin B12 or folic acid deficiency, active bleeding, hemolytic anemia, hematological malignancies, etc.).
* Contraindications and related risks of Roxadustat:
* People who are allergic to roxadustat or any of its excipients.
* Uncontrolled hypertension (sitting systolic blood pressure remains > 160 mmHg or diastolic blood pressure > 100 mmHg after active antihypertensive treatment).
* There have been thrombotic events such as acute myocardial infarction, unstable angina pectoris, stroke, deep vein thrombosis or pulmonary embolism within the past six months.
* Those with known active malignant tumors or undergoing anti-tumor treatment (except for basal cell carcinoma, etc.) are excluded.
* Diseases affecting muscle metabolism and assessment:
* Severe thyroid dysfunction (uncontrolled).
* Diagnosed with chronic liver cirrhosis, acute exacerbation of chronic obstructive pulmonary disease (COPD), congestive heart failure (NYHA class IV), and other chronic diseases that seriously affect muscle metabolism.
* Due to severe limitations in limb movement caused by rheumatoid arthritis, Parkinson's disease, spinal cord injury, etc., it is impossible to complete muscle strength and functional tests.
* Long-term and excessive use of glucocorticoids (equivalent to prednisone > 7.5 mg/day) or other drugs that may affect muscle metabolism (such as androgens).
* Other serious systemic diseases:
* Severe liver dysfunction (Child-Pugh grade C or ALT/AST > 3 times the upper limit of normal).
* Active, uncontrolled severe infection.
* Life expectancy is less than one year.
* Special circumstances related to the research:
* A kidney transplant is planned within the next six months.
* Has participated in any other interventional clinical trials within the past 3 months.
* Poor compliance and special populations:
* There are mental or cognitive impairments, making it impossible to understand or cooperate with the research.
* Pregnant or lactating women, or women of childbearing age who are unwilling to take effective contraceptive measures during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The impacts of different drug therapies (roxadustat or erythropoietin) on the sarcopenia status of patients | 16 weeks
  The risk of sarcopenia in patients was evaluated using the SARC-Calf assessment form.
The impacts of different drug therapies (roxadustat or erythropoietin) on the sarcopenia status of patients | 16 weeks
  Muscle strength was measured by employing a handgrip dynamometer on the dominant hand of the patients.
The impacts of different drug therapies (roxadustat or erythropoietin) on the sarcopenia status of patients | 16 weeks
  The muscle area at the L3 level was assessed via CT scan.
The impacts of different drug therapies (roxadustat or erythropoietin) on the sarcopenia status of patients | 16 weeks
  The locomotor ability of patients was evaluated through the 6-meter walking test.

SECONDARY OUTCOMES:
The impacts of two distinct drug therapies on the amelioration of renal anemia in patients | 16 weeks
  Measurement of hemoglobin (Hb) concentration
The impacts of two distinct drug therapies on the amelioration of renal anemia in patients | 16 weeks
  Measurement of mean corpuscular volume (MCV)
The impacts of two distinct drug therapies on the amelioration of renal anemia in patients | 16 weeks
  Measurement of mean corpuscular hemoglobin (MCH)
The impacts of two distinct drug therapies on the amelioration of renal anemia in patients | 16 weeks
  Measurement of mean corpuscular hemoglobin concentration (MCHC)
The impacts of two distinct drug therapies on the amelioration of renal anemia in patients | 16 weeks
  Measurement of serum iron levels

OTHER OUTCOMES:
The incidences of adverse events in the two groups of patients | 16 weeks
  Blood pressure was self - measured by patients on a daily basis.
The incidences of adverse events in the two groups of patients | 16 weeks
  Patients are required to report any symptomatic discomforts promptly.

REFERENCES:
- [Background] Sekar J, Attaway AH. The intersection of HIF-1alpha, O-GlcNAc, and skeletal muscle loss in chronic obstructive pulmonary disease. Glycobiology. 2023 Dec 25;33(11):873-878. doi: 10.1093/glycob/cwad081. PMID 37812446
- [Background] Yin A, Fu W, Elengickal A, Kim J, Liu Y, Bigot A, Mamchaoui K, Call JA, Yin H. Chronic hypoxia impairs skeletal muscle repair via HIF-2alpha stabilization. J Cachexia Sarcopenia Muscle. 2024 Apr;15(2):631-645. doi: 10.1002/jcsm.13436. Epub 2024 Feb 9. PMID 38333911
- [Background] Cirillo F, Mangiavini L, La Rocca P, Piccoli M, Ghiroldi A, Rota P, Tarantino A, Canciani B, Coviello S, Messina C, Ciconte G, Pappone C, Peretti GM, Anastasia L. Human Sarcopenic Myoblasts Can Be Rescued by Pharmacological Reactivation of HIF-1alpha. Int J Mol Sci. 2022 Jun 26;23(13):7114. doi: 10.3390/ijms23137114. PMID 35806119
- [Background] Liu H, Li Y, Xiong J. The Role of Hypoxia-Inducible Factor-1 Alpha in Renal Disease. Molecules. 2022 Oct 28;27(21):7318. doi: 10.3390/molecules27217318. PMID 36364144